CLINICAL TRIAL: NCT00829647
Title: A Phase I/II Study of Combination Dasatinib and Lenalidomide in Purine Analogue-Failed Chronic Lymphocytic Leukemia
Brief Title: A Study Using Two Oral Chemotherapy Agents for Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: Scripps Health (Other)
Collaborators: Bristol-Myers Squibb (Industry); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Darren Sigal, MD, Principal Investigator, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLL084993
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: CLL; dasatinib; lenalidomide; sprycel; revlimid; CLL relapsed or refractory to fludarabine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Dasatinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- combination dasatinib plus lenalidomide (Experimental): dasatinib 70 mg po daily plus lenalidomide 2.5 md po daily
  Interventions: Drug: dasatinib and lenalidomide

INTERVENTIONS:
Drug: dasatinib and lenalidomide — dasatinib will be started at 70mg/day po and lenalidomide will be started at 2.5mg/day po
  Other Names: spyrcel and revlimid

SUMMARY:
Dasatinib and lenalidomide are both prescribed for use in patients with different cancers of the blood. This study is experimental because neither drug has been approved by the Food and Drug Administration for the treatment of chronic lymphocytic leukemia. There are few standard treatments when fludarabine is no longer effective in patients with CLL. Some patients have received additional combination therapy with fludarabine, Campath, bone marrow transplants or supportive care. Dasatinib and lenalidomide have been effective in high-risk CLL patients in other pilot mono therapy studies. The combination of dasatinib and lenalidomide has not been studied in humans before and this study is designed to test whether this combination is safe to use.

DETAILED DESCRIPTION:
CLL is an incurable disease with current therapies. Modern chemoimmunotherapies, including combinations of rituximab and purine nucleoside analogues (fludarabine, cladribine, and pentostatin), offer the possibility for improved survival, but all patients will eventually relapse. Patients with relapsed or refractory disease will only experience diminishing benefits with additional lines of therapy. In addition, patients with high-risk CLL have poor responses to even first-line therapies. Lenalidomide and dasatinib have non-overlapping proposed mechanisms of action. Single agent phase II studies with lenalidomide and dasatinib have demonstrated responses in heavily pretreated and high-risk patients. For these reasons, we propose to treat patients with relapsed and/or refractory CLL to purine nucleoside analogue therapy with combination lenalidomide and dasatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign a written informed consent including a HIPAA form according to institutional guidelines
2. Age ≥18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Immunophenotypically confirmed diagnosis of B-CLL, who either have Rai stage III/IV disease or require treatment for Rai stage I/II disease as defined by criteria based on the NCI 1996 guidelines (Appendix VII and IX).
5. Relapsed and/or refractory disease to a purine nucleoside analogue (pentostatin, fludarabine, or cladribine). Relapse is defined as a patient who has previously achieved the clinicopathologic criteria for a CR or PR, but after a period of ≥ 6 months demonstrates evidence of disease progression. Refractory is defined as a patient progressing on therapy or who cannot maintain at least a PR for ≥ 6 months (Appendix IV). The patient may have had therapy subsequent to receiving a purine nucleoside analogue, but must also have relapsed or been refractory to this most recent therapy (Appendix IV).
6. ECOG performance status of ≤ 2 at study entry (see Appendix X).
7. Laboratory test results within these ranges:

   * Absolute neutrophil count ≥ 1,000/mm3
   * Platelet count ≥ 50,000/mm³
   * Serum creatinine ≤ 1.5 mg/dL. Subjects with serum creatinine > 1.5 mg/dL may be eligible if they have creatinine clearance of ≥ 60 mL/min by Cockroft-Gault formula.
   * Total bilirubin ≤ 1.5 mg/dL
   * AST (SGOT) and ALT (SGPT) ≤ 2 x ULN or ≤ 5 x ULN if hepatic metastases are present.
8. Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast. Patients with low- and intermediate-risk prostate cancer who have had either local therapy (radiation or surgery) or are actively receiving hormonal therapy will also be allowed. Patients being observed with "watchful waiting" will be excluded. Low- and intermediate-risk prostate cancer will be defined as PSA ≤ 20, Gleason score ≤ 7, and AJCC clinical stage of ≤ T2b.
9. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix I: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND also Appendix II: Education and Counseling Guidance Document.
10. Ability to take oral medication (dasatinib and lenalidomide must be swallowed whole).
11. Concomitant Medications

    * Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib)
    * Bisphosphonate use will be restricted

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide and/or dasatinib)
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide or dasatinib
8. Known positive for HIV or infectious hepatitis, type A, B or C.
9. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness
10. Women who:

    * are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or
    * have a positive pregnancy test at baseline, or
    * are pregnant or breastfeeding
11. Concomitant Medications, any of the following should be considered for exclusion:

    * Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib)
    * quinidine, procainamide, disopyramide
    * amiodarone, sotalol, ibutilide, dofetilide
    * erythromycin, clarithromycin
    * chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
    * cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
12. History of significant bleeding disorder unrelated to cancer, including:

    * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
    * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
    * Ongoing or recent (≤ 3 months) significant bleeding from any cause
13. Cardiac Symptoms; any of the following should be considered for exclusion:

    * Uncontrolled angina, congestive heart failure or MI within (6 months)
    * Diagnosed congenital long QT syndrome
    * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
    * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
    * Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
14. Concurrent medical condition which may increase the risk of toxicity, including:

    • Pleural or pericardial effusion of any grade
15. Evidence of laboratory TLS by Cairo-Bishop criteria (Appendix XIII) (subjects may be enrolled upon correction of electrolyte abnormalities)
16. Patients with an increased risk for thromboembolic events at baseline, including patients with a history of prior thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Safety and maximum tolerated dose (phase I) and overall response rate (phase II) | 6 months

SECONDARY OUTCOMES:
Assess responses in subgroups of high-risk patients, including 17p- and 11q- deletion, and CD38 and ZAP-70 positive expression | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Darren Sigal, MD, Principal Investigator — Staff Scripps Cancer Center

IPD SHARING:
Plan to Share IPD: No
There is no data to share.

REFERENCES:
- [Background] Chanan-Khan A, Miller KC, Musial L, Lawrence D, Padmanabhan S, Takeshita K, Porter CW, Goodrich DW, Bernstein ZP, Wallace P, Spaner D, Mohr A, Byrne C, Hernandez-Ilizaliturri F, Chrystal C, Starostik P, Czuczman MS. Clinical efficacy of lenalidomide in patients with relapsed or refractory chronic lymphocytic leukemia: results of a phase II study. J Clin Oncol. 2006 Dec 1;24(34):5343-9. doi: 10.1200/JCO.2005.05.0401. Epub 2006 Nov 6. PMID 17088571
- [Background] Ferrajoli A, Lee BN, Schlette EJ, O'Brien SM, Gao H, Wen S, Wierda WG, Estrov Z, Faderl S, Cohen EN, Li C, Reuben JM, Keating MJ. Lenalidomide induces complete and partial remissions in patients with relapsed and refractory chronic lymphocytic leukemia. Blood. 2008 Jun 1;111(11):5291-7. doi: 10.1182/blood-2007-12-130120. Epub 2008 Mar 11. PMID 18334676